CLINICAL TRIAL: NCT00945555
Title: Multi-Center, Non-Interventional, Observational Study To Evaluate The Antibacterial Therapeutical Options In Febrile Neutropenia Patients
Brief Title: Observational Non-Interventional Study Of Febrile Neutropenia Patients To Evaluate Antibacterial Therapeutical Options
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1891006
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Febrile Neutropenia
Keywords: Antibacterials; Classification of antibacterial agent; Febrile neutropenia; Turkey
MeSH Terms: conditions — Febrile Neutropenia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Participants with febrile neutropenia who received antibacterial treatment per investigator's judgment
  Interventions: Drug: Antibacterial agent for the treatment of febrile neutropenia

INTERVENTIONS:
Drug: Antibacterial agent for the treatment of febrile neutropenia — The antibacterial agent used by the investigators for febrile neutropenia will be determined and classified in the preference order

SUMMARY:
The purpose of this study was to define and classify antibacterial agents used in Turkey for patients with febrile neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years old and above.
* Patients who have undergone allogeneic/autologous or peripheral stem cell transplantation following induction or consolidation treatment due to acute hematological malignancy.
* Patients who have a neutrophil count below 500 cells per cubic millimeter (cells/mm^3) or below 1000 cells/mm^3 with an expectancy to rapidly decrease below 500 cells/mm^3.
* Patients with a body temperature more than or equal to (≥)38.3 degrees Celsius (101 degrees Fahrenheit) on single oral measurement or detected ≥38.0 degrees Celsius for at least an hour and thus started on antibacterial treatment will be included in the trial.

Exclusion Criteria:

- Patients who are pregnant or considering pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with febrile neutropenia who were planning to take antibacterial treatment.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Turkey (Türkiye) (5):
  - Pfizer Investigational Site, Kayseri, Turkey
  - Pfizer Investigational Site, Kocaeli, Turkey
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Bursa
  - Pfizer Investigational Site, Istanbul

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants with febrile neutropenia who received treatment as determined by the physician
Period: Overall Study
Arm/Group | All Participants
Started | 264
Completed | 236
Not Completed | 28
Not completed — Referred to another hospital | 5
Not completed — Worsening condition, intensive care unit | 1
Not completed — Withdrawal by Subject | 2
Not completed — Participant continued treatment at home | 1
Not completed — Death | 18
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.41 (16.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 168

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Receiving Antibacterial Agents Preferred by the Turkish Centers Monitoring Febrile Neutropenia (FEN) in Their Therapeutical Approach: Empirical
Time Frame: Baseline
Population: All participants enrolled in the study. Participants may be counted more than once because they may have received more than one antibacterial agent.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 264
percentage of participants
  Cefoperazone/Sulbactam (S) | 33.3
  Piperacillin-Tazobactam (P) | 32.6
  Imipenem+Cilastatin Sodium (I) | 26.1
  Meropenem (M) | 8.0
  I+Vancomycin | 3.0
  I+Teicoplanin | 3.0
  Ceftazidime | 2.7
  S+Teicoplanin | 1.5
  P+Teicoplanin | 1.5
  M+Vancomycin | 1.1
  P+Moxifloxacin | 0.8
  M+Teicoplanin | 0.8
  M+S+Teicoplanin | 0.8
  P+I | 0.8
  Teicoplanin+Ceftazidime | 0.4
  P+Vancomycin | 0.4
  P+Clarithromycin | 0.4
  M+S+Trimethoprim-Sulfamethoxazole | 0.4
  M+S+ Teicoplanin+Ofloxacin | 0.4
  M+S+ Teicoplanin+Colistin Sulfate | 0.4
  M+S | 0.4
  I+Teicoplanin+Moxifloxacin | 0.4
  I+S | 0.4
  I+P+Teicoplanin | 0.4
  I+M+S | 0.4
  I+M | 0.4
  I+Linezolid | 0.4

2. Primary Outcome: Percentage of Participants Receiving Antibacterial Agents Preferred by the Turkish Centers Monitoring FEN in Their Therapeutical Approach: Targeted
Time Frame: Baseline
Population: All participants enrolled in the study who received treatment for febrile neutropenia. Number of participants analyzed=number of participants who received an antibacterial drug for the treatment of febrile neutropenia. Participants may be counted more than once because they may have received more than one antibacterial agent.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 259
percentage of participants
  Imipenem+Cilastatin Sodium (I) | 34.7
  Cefoperazone/Sulbactam (S) | 29.0
  Piperacillin-Tazobactam (P) | 27.8
  Meropenem (M) | 12.4
  I+Teicoplanin (T) | 5.8
  P+T | 3.9
  S+T | 3.9
  I+Vancomycin | 2.7
  Ceftazidime | 2.3
  P+Vancomycin | 1.9
  M+T | 1.5
  M+Vancomycin | 1.5
  T | 1.2
  I+Fluconazole (F) | 0.8
  I+Linezolid (L) | 0.8
  M+S+T | 0.8
  P+Moxifloxacin | 0.8
  F+I+Vancomycin | 0.4
  I+Amikacin | 0.4
  I+Ganciclovir | 0.4
  I+Metronidazole | 0.4
  I+Ceftazidime | 0.4
  I+Ceftriaxone | 0.4
  I+Ciprofloxacin+Tigecycline | 0.4
  I+T+Amikacin | 0.4
  I+T+F | 0.4
  I+T+Moxifloxacin | 0.4
  I+Voriconazole (V)+T+Ciprofloxacin+Caspofungin | 0.4
  L+M+I+Zanamivir | 0.4
  M+I | 0.4
  M+I+Ceftriaxone | 0.4
  M+I+T | 0.4
  M+L | 0.4
  M+S+I | 0.4
  M+S+L+T | 0.4
  M+S+T+Metronidazole | 0.4
  M+S+T+Ofloxacin | 0.4
  M+S+Trimethoprim-Sulfamethoxazole (Trimet-Sulfa) | 0.4
  M+T+F+Caspofungin acetate | 0.4
  M+T+Caspofungin acetate | 0.4
  M+T+Ofloxacin | 0.4
  M+T+Trimet-Sulfa | 0.4
  M+V | 0.4
  P+I | 0.4
  P+I+F | 0.4
  P+I+Vancomycin | 0.4
  P+Colistin | 0.4
  P+Levofloxacin | 0.4
  P+Metronidazole | 0.4
  S+I | 0.4
  S+I+L+Amphotericin | 0.4
  S+I+L+Ciprofloxacin+Trimet-Sulfa+Amphotericin | 0.4
  S+I+L+V+Clarithromycin | 0.4
  S+I+V+T | 0.4
  S+L+T | 0.4
  S+M+L+V+T+Trimet-Sulfa+Amphotericin | 0.4
  S+Ciprofloxacin+Acyclovir | 0.4
  S+T+Acyclovir | 0.4
  S+Valaciclovir | 0.4
  T+Ceftazidime | 0.4
  T+Valaciclovir | 0.4
  V+M+S+T+Valaciclovir | 0.4

3. Secondary Outcome: Mean Body Temperature
Time Frame: Baseline, Day 4, Day 7 on Average (till the End of Treatment)
Population: All participants enrolled in the study. n=number of participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | All Participants
Number analyzed (Participants) | 264
Degree Celsius
  Baseline (n=264) | 38.5 (0.4)
  Day 4 (n=261) | 37.4 (0.9)
  Day 7 on Average (End of Treatment) (n=257) | 36.7 (0.6)

4. Secondary Outcome: Mean Neutrophil Count
Time Frame: Baseline, Day 4, Day 7 on Average (till the End of Treatment)
Population: All participants enrolled in the study. Number of participants analyzed=number of participants with available data. n=number of participants with data available at that time point.
Measure: Mean (Standard Deviation); unit: neutrophils per cubic millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 254
neutrophils per cubic millimeter
  Baseline (n=254) | 220.1 (997.2)
  Day 4 (n=239) | 394.8 (2204.7)
  Day 7 on Average (End of Treatment) (n=242) | 1222.1 (3860.3)

5. Secondary Outcome: Percentage of Participants in Whom New Infection Was Determined on Day 4
Time Frame: Day 4
Population: All participants enrolled in the study. Number of participants analyzed=participants with new infection diagnosed on Day 4.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
percentage of participants
  Primary bloodstream infection | 15.5
  Bloodstream infection originating from catheter | 14.1
  Urinary tract infection | 11.3
  Catheter infection | 11.3
  Mucositis | 9.9
  Fungal pneumonia | 8.5
  Fungal infection in the lung | 7.0
  Bacteriemia | 7.0
  Oral candidiasis | 4.2
  Pneumonia | 4.2
  Oral mucositis | 4.2
  Dental abscess | 2.8
  Herpes labialis | 2.8
  Diarrhea | 2.8
  Cellulitis | 2.8
  Influenza | 2.8
  Bronchoalveolar lavage (BAL) legionella | 1.4
  BAL Chlamydia Pneumonia | 1.4
  Cytomegalovirus (CMV) infection | 1.4
  Deep vein thrombosis+thrombophlebitis | 1.4
  Diabetic foot infection | 1.4
  Fever of unknown origin | 1.4
  Cellulitis gluteal region | 1.4
  H1N1 | 1.4
  Intra-abdominal infection | 1.4
  Candidemia | 1.4
  Catheter entry infection | 1.4
  Oral fungal infection | 1.4
  Esophagitis | 1.4
  Consolidation in left lung upper zone | 1.4
  Typhlitis | 1.4
  Tunnel infection | 1.4
  Tracheal aspiration | 1.4

6. Secondary Outcome: Percentage of Participants in Whom New Infection Was Determined at End of Treatment
Time Frame: Day 7 on Average (till the End of Treatment)
Population: All participants enrolled in the study. Number of participants analyzed = number of participants with new infection diagnosed at end of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 59
percentage of participants
  Catheter infection | 23.7
  Bacteriemia | 13.6
  Pneumonia | 8.5
  Primary bloodstream infection | 6.8
  Soft tissue infection | 5.1
  Typhilitis | 5.1
  Urinary tract infection | 5.1
  Fungal pneumonia | 5.1
  Abscess | 5.1
  Fungal infection in lung | 5.1
  Sinusitis | 3.4
  Sepsis | 3.4
  Mucositis | 3.4
  Influenza | 3.4
  Fever of unknown origin | 3.4
  Anal fissure+hemorrhoid | 3.4
  Bloodstream infection originating from catheter | 3.4
  Tunnel infection | 1.7
  Subdural-intradural hematoma abscess | 1.7
  Pneumocystis pneumonia | 1.7
  Orofaringeal candidiasis | 1.7
  Intra abdominal infection | 1.7
  Herpes labialis | 1.7
  Vancomycin-resistant enterococci in stool | 1.7
  Gastroenteritis | 1.7
  Fusariosis (skin+eye) | 1.7
  BAL pseudomonas aspergillosa | 1.7
  Diphtheroid bacillus in 2 blood cultures | 1.7

7. Secondary Outcome: Percentage Survivors
Time Frame: Day 7 on Average (till the End of Treatment)
Population: All participants enrolled in the study. Number of participants analyzed=number of participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 256
percentage of participants | 93.0

8. Secondary Outcome: Percentage of Participants Who Had a Treatment Modification
Time Frame: Day 4, Day 7 on Average (till the End of Treatment)
Population: All participants enrolled in the study. Number of participants analyzed=number of participants who had a treatment modification at any time point. n=number of participants who had data available at that specific time point.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 258
percentage of participants
  Day 4 (n=258) | 24.8
  Day 7 on Average (End of Treatment) (n=253) | 50.6

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/264
Other Adverse Events (participants affected / at risk) | 19/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=264)
Chilling, shivering, fever reaction (General disorders) | 1
Systemic allergic reaction-hypotension (General disorders) | 1
Diarrhea (General disorders) | 1
Hepatotoxicity (General disorders) | 1
Elevation of creatinine level (General disorders) | 1
Elevation of transaminase (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=264)
Diarrhea (General disorders) | 2 (2)
Hepatotoxicity (General disorders) | 1 (1)
Mucositis (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Nausea, vomiting (General disorders) | 6 (7)
Nephrotoxicity (General disorders) | 1 (1)
Rash (General disorders) | 8 (9)
Vomiting-headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.